CLINICAL TRIAL: NCT02152917
Title: Comparison of Floseal® and Tranexamic Acid on Bleeding Control After Total Knee Arthroplasty - Randomized Prospective Study
Brief Title: Comparison of Floseal® and Tranexamic Acid on Bleeding Control After Total Knee Arthroplasty
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Marco Kawamura Demange, Assistant Professor, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014/11297
Record Dates: First submitted 2014-05-29; First posted 2014-06-02 (Estimated); Last update posted 2014-06-02 (Estimated); Status verified 2014-05

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Tranexamic Acid; FloSeal Matrix

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Tranexamic acid (Active Comparator): A dose of tranexamic acid (10mg/Kg) will be administered 20 minutes before inflating the pneumatic tourniquet and another dose 15 minutes after the tourniquet release.
  Interventions: Drug: Tranexamic acid
- Floseal® (Active Comparator): Floseal® will be applied in regions of potential bleeding before the release of the pneumatic tourniquet.
  Interventions: Drug: Floseal®
- Control group (No Intervention)

INTERVENTIONS:
Drug: Tranexamic acid
  Other Names: TA
  Arms: Tranexamic acid
Drug: Floseal®
  Arms: Floseal®

SUMMARY:
The total knee arthroplasty (TKA) is a well established option for the treatment of osteoarthritis in this joint. Nevertheless, there are still some concerns related to the peri-operative management of elderly patients, highlighting the complications related to medical comorbidity and bleeding produced by surgery. One of the proposed methods to decrease postoperative bleeding, which has been accumulating favorable evidence, is the use of tranexamic acid (TA). Several studies (including prospective randomized trials with placebo group) showed excellent results with TA intravenous administration during TKA, reducing the amount of bleeding, the drop in hemoglobin and the need for blood transfusion. Another alternative to minimize bleeding is the use of topical hemostatic agent Floseal®, composed of thrombin and bovine gelatin. This substance has presented significant benefits on bleeding control in several areas of medicine, including orthopedic surgery, but no action has yet been established in TKA. The main objective is to evaluate the amount of bleeding, the drop in hemoglobin and the need for blood transfusion after TKA, comparing the use of TA, Floseal® and a control group. The secondary objective is to evaluate the rate of adverse events in the studied groups.

ELIGIBILITY:
Inclusion Criteria:

* Indication for total knee arthroplasty
* No previous knee surgery
* Absence of inflammatory arthritis
* Absence of stiff knee
* Absence of the following factors: renal failure, liver failure, severe heart failure, respiratory failure, history of thromboembolic events, bleeding disorders, previous strokes

Exclusion Criteria:

* None

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2014-02; Primary Completion 2015-02 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
Amount of bleeding | First two days post-operative
  Measure of the drain volume on the first two days post-operative
Drop in hemoglobin | Three days postoperative
  Difference between the preoperative hemoglobin and hemoglobin in the third postoperative

SECONDARY OUTCOMES:
Adverse events | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Camilo P Helito, M.D., Principal Investigator — University of Sao Paulo; Ricardo G Gobbi, M.D., Principal Investigator — University of Sao Paulo; Luis Eduardo P Tirico, M.D., Principal Investigator — University of Sao Paulo; Marco K Demange, Ph.D., Principal Investigator — University of Sao Paulo; Jose R Pecora, Ph.D., Study Director — University of Sao Paulo; Gilberto L Camanho, Ph.D., Study Chair — University of Sao Paulo; Marcelo B Bonadio, M.D., Principal Investigator — University of Sao Paulo
Locations (1):
- Hospital das Clinicas - University of Sao Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Helito CP, Bonadio MB, Sobrado MF, Giglio PN, Pecora JR, Camanho GL, Demange MK. Comparison of Floseal(R) and Tranexamic Acid for Bleeding Control after Total Knee Arthroplasty: a Prospective Randomized Study. Clinics (Sao Paulo). 2019 Nov 25;74:e1186. doi: 10.6061/clinics/2019/e1186. eCollection 2019. PMID 31778430